CLINICAL TRIAL: NCT05955287
Title: A Pilot Study to Determine the Feasibility of a Couples' Oriented Intervention to Promote CPAP Adherence Among African American Patients With Obstructive Sleep Apnea
Brief Title: CPAP Adherence Pilot Study Among African Americans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Daryl Thornton, MD, Co-Director, Center for Reducing Health Disparities Co-Director of Education, Population Health Research Institute Director, Medical Intensive Care Unit Associate Professor, Department of Internal Medicine, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000055
Record Dates: First submitted 2023-02-02; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Sleep Apnea
Keywords: obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: In the intervention group, patients with OSA and their bed partners will participate in two 1-hour video support groups at 2 weeks and 2 months ran by patients with OSA and their bed partners. Patients with OSA and their bed partners will be contacted in their preferred manner (text messages, email, or phone call) periodically (no more than 4 per week) to determine how well they slept, to encourage them to use their CPAP, or to remind them to contact study staff if they are having difficulty using their CPAP.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couple Intervention (Experimental): Patients will receive usual care. In addition, they will participate in virtual OSA support groups led by an African American peer-motivator patient with long-standing OSA and their bed partner. Peer-motivator couples will be trained and certified as competent prior to interacting with study participants. They will share their experiences with managing OSA including coping strategies to maximize CPAP adherence.
  Telemonitoring. Patients and bed partners will receive text messages encouraging CPAP adherence.
  Interventions: Behavioral: Telemonitoring; Behavioral: Peer Based; Behavioral: CPAP Education; Behavioral: Usual Care
- Control (Active Comparator): Patients with CPAP technical difficulties will be encouraged to contact the sleep technologist for assistance. Patients will also attend a 90-minute virtual webinar and question-answer session on hypertension management (1 month), cancer screening (3 months), and weight management (6 months) led by African American physicians with expertise in each topic.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Telemonitoring — Text messages of encouragement will be sent to patients and partners. No more than 2 messages will be sent per week to prevent respondent fatigue.
  Arms: Couple Intervention
Behavioral: Peer Based — Patients and partners will attend OSA virtual support groups led by an African American patient with long-standing OSA and their bed partner. Peer-motivator couples will be trained and certified as competent prior to interacting with study participants. They will share their experiences with managing OSA including coping strategies to maximize CPAP adherence.
  Arms: Couple Intervention
Behavioral: CPAP Education — Patients with OSA and their bed partners will participate in two 1-hour video support groups at 2 weeks and 2 months ran by patients with OSA and their bed partners
  Arms: Couple Intervention
Behavioral: Usual Care — Participants will receive OSA education and CPAP training from providers trained in OSA management.

SUMMARY:
The goal of the study is to determine the feasibility of a behavioral intervention to improve CPAP adherence among African American patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
The Investigators propose to pilot test a couple-oriented intervention in a randomized controlled trial of 20 African American patients diagnosed with moderate to severe OSA and their partners. Half of the patients will receive optimal usual care currently implemented at MetroHealth, consisting of sleep therapist-initiated standardized education about OSA, sleep hygiene, and CPAP use; personalized mask fittings; and follow-up at 1 week to troubleshoot problems with CPAP utilization. Participants will follow up with their sleep providers per usual. The remaining patients and their bed partners will receive a couple-oriented intervention consisting of guideline-recommended best practices for improving CPAP adherence consisting of sleep therapist-initiated standardized education for couples about OSA, sleep hygiene, and CPAP use; personalized mask fittings; and follow-up at 1 week to troubleshoot problems with CPAP utilization. Couples will participate in two couple-oriented support groups led by an African American patient with long standing OSA treated with CPAP and their partner. Patients and partners will receive tailored text messages encouraging adherence. In addition, couples will receive five 60-minute virtual cognitive behavioral couple therapy sessions with a health psychologist trained in behavioral sleep medicine that will focus on enhancing couples' knowledge of CPAP, patients' self-efficacy to use CPAP, couple's relationship dynamics, and partners' skill and self-efficacy in assisting the patient with CPAP adherence.

ELIGIBILITY:
Inclusion Criteria:

* Must have same bed partner(s) for at least 6 months.
* Must be at least 18 years of age

Exclusion Criteria:

* Must be Proficient in speaking English
* Non-compliance to management of OSA
* Apnea hypopnea Index ≥ 15 events/hours
* Terminally ill
* Mentally incompetent
* unstable housing
* need for BPAP or VPAP\PAP).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
CPAP Adherence | 3 months
  Mean hours per night of CPAP use

SECONDARY OUTCOMES:
Sleep Apnea Quality of Life | 3 months
  Calgary Sleep Apnea Quality of Life Index. 84 items with higher scores suggesting higher quality of life
Patient and Partner Sleepiness | 3 months
  Epworth Sleepiness Scale (ESS) - 8 items, with scoring range 0 - 24. Higher scores are associated with increased sleepiness.
Patient and Partner Quality of Sleep | 3 months
  Functional Outcomes of Sleep Questionnaire (FOSQ-10) Patient and Partner Functional Status assessed in 10 questions with lower scores suggesting worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: John D Thornton, MD, MPH, Principal Investigator — MetroHealth System, Ohio
Locations (1):
- MetroHealth Medical System, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Results from the study will be shared through the publication of findings in research journals and via presentation at scientific meetings. Results will be directly shared with participants upon inquiry.

DOCUMENTS (1):
  • Study Protocol (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT05955287/Prot_000.pdf